CLINICAL TRIAL: NCT02224950
Title: Study to Examine the Benefits of Fabric Made With Lyocell/Chitosan/Ceramide in the Treatment of Children With Mild to Moderate Eczema
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Withdrawn from IRB before approval
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UofMLyocell
Record Dates: First submitted 2014-08-21; First posted 2014-08-25 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Atopic Dermatitis
Keywords: Atopic dermatitis; eczema; alternative therapy; complementary therapy; moisturizer
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Placebo Comparator): Non-medicated Emollient with no Clothing Covering Upper Limb - "Baseline/Control" Cells
  Interventions: Device: Non-medicated Emollient plus Lyocell/Chitosan Sleeve
- Sleeve 2 (Active Comparator): Non-medicated Emollient plus Lyocell/Chitosan Sleeve
  Interventions: Other: Non-medicated Emollient plus Cotton Sleeve
- Placebo Sleeve (Placebo Comparator): Non-medicated Emollient plus Cotton Sleeve
  Interventions: Other: Placebo Sleeve

INTERVENTIONS:
Device: Non-medicated Emollient plus Lyocell/Chitosan Sleeve
  Arms: Control
Other: Non-medicated Emollient plus Cotton Sleeve
  Arms: Sleeve 2
Other: Placebo Sleeve
  Arms: Placebo Sleeve

SUMMARY:
The study will primarily focus on evaluating the benefits of using a lyocell/chitosan/ceramide fabric as a treatment for young children with mild or moderate eczema. More specifically, the study will focus on the upper limb area in these patients and will examine whether wearing a sleeve made from a lyocell/chitosan/ceramide fabric can improve eczema symptoms compared with wearing a cotton sleeve, no sleeve, or the lyocell / chitosan combination. Patients will be evaluated at 3 intervals over a 3-week period using the following four variables: an eczema severity index, amount of itching, bacteria levels in the affected areas of skin, and amount of water loss in the affected areas.

DETAILED DESCRIPTION:
The study will be evaluated using the following four variables: an eczema severity index, amount/severity of itching, bacteria levels in the affected areas of skin, and amount of water loss in the affected areas. The eczema severity will be scored using the EASI (upper limb subscale); itch will be assessed with a Visual Analog Scale for itch; the skin will be swabbed for bacterial cultures and results are quantified based on microbiology lab standards to be mild, moderate or heavy growth of the bacteria identified; and transepidermal water loss (TEWL) will be measured using a tewameter/capacitive moisture sensor.

ELIGIBILITY:
Inclusion Criteria:

* Age 3 months to 5 years
* Mild or moderate atopic dermatitis, as determined by Investigator Global Assessment Criteria

Exclusion Criteria:

* Non-English speaking subjects/families
* Families unable to complete study requirements

Ages: 3 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2014-11; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Benefit of ceramide embedded fabric | 3 weeks
  Whether wearing a sleeve made from a lyocell/chitosan/ceramide fabric can improve eczema symptoms compared to wearing a cotton sleeve, no sleeve, or the lyocell / chitosan combination.

SECONDARY OUTCOMES:
Bacterial growth | 3 weeks
  Is bacterial growth affected by the fabric combination?

OTHER OUTCOMES:
Trans-epidermal water loss | 3 weeks
  Is trans-epidermal water loss affected by the fabric combination?

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Hook, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States